CLINICAL TRIAL: NCT03787017
Title: A Randomized, Open-label, Single-dosing, 2X2 Crossover Study to Compare the Safety and Pharmacokinetics of FDC of MP-513 20mg and Metformin XR 1000mg With Coadministration of the Two Separate Drugs in Healthy Male Volunteers
Brief Title: A Study to Compare MP-513 20mg & Metformin XR 1000mg FDC With Coadministration of the Two Separate Drugs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MP_C101
Record Dates: First submitted 2015-10-05; First posted 2018-12-26 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Metformin

ARMS (2):
- Sequence Group A (Experimental): 1. 1st period : coadministration of 1 tablet of MP-513 20mg and 1 tablet of Metformin XR 1000mg, single-dose under fasted
  2. 2nd period : 1 tablet of FDC(MP-513 20mg/Metformin XR 1000mg), single-dose under fasted
  Interventions: Drug: FDC(MP-513 20mg/Metformin XR 1000mg); Drug: MP-513 20mg; Drug: Metformin XR 1000mg
- Sequence Group B (Experimental): 1. 1st period : 1 tablet of FDC(MP-513 20mg/Metformin XR 1000mg), single-dose under fasted
  2. 2nd period : coadministration of 1 tablet of MP-513 20mg and 1 tablet of Metformin XR 1000mg, single-dose under fasted
  Interventions: Drug: FDC(MP-513 20mg/Metformin XR 1000mg); Drug: MP-513 20mg; Drug: Metformin XR 1000mg

INTERVENTIONS:
Drug: FDC(MP-513 20mg/Metformin XR 1000mg)
  Other Names: HL1351
Drug: MP-513 20mg
  Other Names: Tenelia 20mg
Drug: Metformin XR 1000mg
  Other Names: Glucophage XR 1000mg

SUMMARY:
The purpose of this study is to compare the safety and pharmacokinetic characteristics of fixed-dose combination of MP-513 20mg and Metformin XR 1000mg with coadministration of the two separate drugs in healthy male volunteers.

DETAILED DESCRIPTION:
1. Randomized, Open-label, Single-dosing, Two-treatment, Two-sequence, Two-period, crossover design
2. Wash-out period : 14days from the first dosing
3. Drug concentration analytical device : UPLC-MS/MS

ELIGIBILITY:
Inclusion Criteria:

* A healthy male adult at the age of 20 to 45 (both inclusive) at the time of screening test.
* Body weight equal to or greater than 55 kg and calculated ideal body weight (IBW) within ±20%
* An individual who has been given and fully understood detailed explanations about this study, decides to participate in the study of his own will, and provides written informed consent to comply with instructions.

Exclusion Criteria:

* History or presence of any clinically significant diseases in the hepatobiliary, renal, nervous(central or peripheral), respiratory, hemato-oncology, cardiovascular, urinary, musculoskeletal, immune, ear, nose and throat (ENT), mental, and, particularly, endocrine systems (e.g., diabetes mellitus, hyperlipidemia, etc.).
* History of any gastrointestinal disease that may affect absorption of the study drug (Crohn's disease, ulcer, acute or chronic pancreatitis, etc.) or gastrointestinal surgeries (except for simple appendectomy or hernia repair).
* Hypersensitivity to MP-513 or drugs containing metformin or other drugs in the same class as ingredients or to other drugs
* Vital signs in a sitting position corresponding to at least one of the following criteria: systolic blood pressure ≥ 140 mmHg or < 90 mmHg, or diastolic blood pressure ≥ 95 mmHg or < 60mmHg.
* Serum creatine > upper limit of reference range
* Required to refrain from food intake for at least 24 hours during the study period due to surgery or religious reason.
* History or presence of drug abuse.
* Administration of drugs that either induce or inhibit drug metabolizing enzymes, such as barbitals, within 1 month prior to the first dosing.
* Intake of food or beverage containing grapefruit or cranberry within 1 week prior to the first dosing.
* Administration of any ethical drugs or traditional Korean herbal medicines within 2 weeks or any over-the-counter drugs or vitamin products within 1 week prior to the first dosing
* An individual who participated in another clinical trial and was administered any investigational product within 2 months prior to the first dosing.
* Whole blood donation within 2 months, apheresis donation within 1 month, or blood transfusion within 1 month prior to the first dosing.
* An individual who drinks excessive amounts of alcohol (more than 21 units/week, 1 unit =10 g of pure alcohol) or who cannot stop drinking alcohol from 24 hours prior to hospital admission through to hospital discharge.
* Having smoked 10 cigarettes/day or more on average over the past 3 months.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
AUC of MP-513 and metformin | - 0(pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hours post-dose(a total of 36 times, with 18 times per period)
  PK assessment
Cmax of MP-513 and metformin | - 0(pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hours post-dose(a total of 36 times, with 18 times per period)
  PK assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical trials center of Chungnam National University Hospital, Daejeon, Jung-gu, South Korea